CLINICAL TRIAL: NCT00845754
Title: Effects of Ketorolac on Post-Operative Febrile Morbidity and Pain Management in Abdominal Myomectomy Patients
Brief Title: Post-Operative Treatment With Ketorolac After Abdominal Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascher-Walsh, Charles, M.D. (Individual)
Collaborators: New York Presbyterian Hospital (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Charles Ascher-Walsh MD, Mount Sinai School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ASW 124
Record Dates: First submitted 2009-02-14; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Febrile Morbidity; Pain
Keywords: Post-operative febrile morbidity; Post-operative pain management
MeSH Terms: conditions — Pain | interventions — Ketorolac; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: saline
- 2 (Active Comparator): Ketorolac
  Interventions: Drug: ketorolac

INTERVENTIONS:
Drug: ketorolac — 15mg IV every6 hours for 4doses
  Other Names: Toradol
  Arms: 2
Drug: saline — 15mg IV every 6hrs for 4 doses
  Arms: 1

SUMMARY:
The purpose of this study is to determine if ketorolac, given after abdominal myomectomy, will decrease the frequency of post-oerative fevers as well as improve post-operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Ant patient undregoing abdominal myomectomy

Exclusion Criteria:

* Patients with contraindication to NSAIDs including history of peptic ulcer disease, renal disease, bleeding diathesis, or hypersensitivity to NSAIDS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 1999-09; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Post-operative febrile morbidity | Inital 24hrs post-operative

SECONDARY OUTCOMES:
Post-operative pain management | Initial 24hrs post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States